CLINICAL TRIAL: NCT02607293
Title: An Exploratory Study to Explore the Correlation Between the Symptoms and Signs of Polycystic Ovarian Syndrome (PCOS) and Risk of Over-response Using New Gonal-f® Pen in Assisted Reproductive Technology (ART) Treatment in China
Brief Title: A Study to Explore Correlation Between Symptoms and Signs of Polycystic Ovarian Syndrome (PCOS) and Risk of Over-response to Ovarian Stimulation
Acronym: ARTIST
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Co., Ltd., China (Industry)
Responsible Party: Sponsor
Other Study IDs: 700623_547
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Gonadotropin releasing hormone agonist (GnRH-a); Gonal-f; Assisted Reproductive Technology
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — follitropin alfa; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Subjects undergoing ART treatment with long GnRH-a or GnRH-ant: Subjects undergoing ART treatment with long GnRH-a protocol or GnRH-ant protocol + Gn + human chorionic gonadotropin (hCG) as per routine clinical practice. No visits or intervention(s) additional to the routine practice of the Investigators will be performed during this observational study.
  Interventions: Drug: Gonal-f®; Drug: Long GnRH agonist; Drug: GnRH antagonist

INTERVENTIONS:
Drug: Gonal-f® — Recombinant human follicle stimulating hormone (r-FSH) will be administered subcutaneously (SC) for about 10 to 20 days along with the ART regimen as routinely practiced by Investigators and according to licensed summary of product characteristics (SmPC label) for the ovarian stimulation.
  Other Names: Recombinant human follicle stimulating hormone
Drug: Long GnRH agonist — As a part of the ART regimen GnRH-agonist will be administered for about 14 to 20 days until down regulation is satisfied as judged by investigator.
Drug: GnRH antagonist — As a part of ART regimen GnRH-antagonist will be initiated and regimen will be as routinely practiced by Investigators and according to licensed SmPC label.

SUMMARY:
This is a Phase IV, prospective, observational, single arm, multicenter trial to identify the population at high risk of overstimulation associated with signs and symptoms of PCOS and examines the utility of 12.5 international units (IU) increment of Gonal-f® new pen for individualized controlled ovarian stimulation (iCOS).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged 20 to 35 years (including both)
* Subjects undergoing ART treatment with long GnRH-a protocol or GnRH-ant protocol + Gn + human chorionic gonadotropin (hCG)
* Subject from whom a written informed consent has been obtained with the understanding that the subject may withdraw consent at any time without prejudice to future medical care

Exclusion Criteria:

* Subjects undergoing ART treatment with mild stimulation protocol
* Concomitant use of Gonal-f® with clomiphene citrate
* With an In vitro fertilisation (IVF)/ Intracytoplasmic sperm injection (ICSI) history of greater than or equal to (>=) 3 times
* Known history of poor ovarian response in a previous COS cycle for IVF/ICSI, defined as less than 4 oocytes retrieved or history of previous cycle cancellation prior to oocyte retrieval due to poor response or poor ovarian reserve, such as Antral follicle count (AFC) less than (<) 5 to 7
* Presence of confirmed or suspected endometriosis Grade III - IV
* Presence of unilateral or bilateral hydrosalpinx
* Using other Gn during stimulation period (such as urinary FSH/human menopausal Gn, except for recombinant luteinizing hormone (r-LH))
* Known history of recurrent miscarriage
* Any contradiction to Gn/GnRH analogues
* Any major systemic disease that as per Investigator's discretion precludes subject for participation in the study
* According to the judgment of the Investigator, any medical condition or any concomitant
* surgery/ medications that would interfere with evaluation of study medications
* Simultaneous participation in another clinical study

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women undergoing ART treatment with long GnRH-a protocol or GnRH-ant protocol using Gonal-f® new pen who are expected to be normal or high responders.
Sampling Method: Non-Probability Sample
Enrollment: 1064 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2017-03-16 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Number of subjects with polycystic ovary | Baseline
Serum Testosterone levels | Baseline
Number of subjects with history of menstrual disorders | Baseline
Number of subjects with hirsutism | Baseline
Number of oocytes retrieved | Baseline up to 2-7 days until end of stimulation cycle (approximately 28 days)

SECONDARY OUTCOMES:
Total Dose of Recombinant Follicle Stimulating Hormone (r-FSH) | Baseline up to 1 month
Daily Dose of Recombinant Follicle Stimulating Hormone (r-FSH) | Baseline up to 1 month
Number of Metaphase II (M II) oocyte retrieved | Baseline up to 2-7 days until end of stimulation cycle (approximately 28 days)
Biochemical pregnancy rate | 4 to 6 Weeks after Embryo transfer (Up to 4 months)
  Biochemical pregnancy was defined as a positive pregnancy test (serum beta-hCG test) of the post-treatment assessment period
Clinical pregnancy rate | 4 to 6 Weeks after Embryo transfer (Up to 4 months)
  Clinical pregnancy was defined as existence of at least one ultrasonography confirmed gestational sac in the uterus, with or without heartbeat.
Implantation Rate | 4 to 6 Weeks after Embryo transfer (Up to 4 months)
  Implantation rate was measured as the number of gestational sacs observed, divided by the number of embryos transferred multiplied by 100.
Number of Subjects With Ovarian Hyper Stimulation Syndrome (OHSS) | Baseline up to 13 month
  OHSS is a syndrome which can manifest with enlarged ovaries, advanced ascites with increased vascular permeability, pleural fluid accumulation, haemoconcentration, and increased blood clotting.
Number of Cycles Cancelled Due to Risk of Ovarian Hyper Stimulation Syndrome (OHSS) | Baseline up to 13 month
  OHSS is a syndrome which can manifest with enlarged ovaries, advanced ascites with increased vascular permeability, pleural fluid accumulation, haemoconcentration, and increased blood clotting.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Co., Ltd., China
Locations (1):
- Merck KGaA Communication Center, Darmstadt, Germany